CLINICAL TRIAL: NCT04636060
Title: Single Center Clinical Trial to Evaluate the Effectiveness of Low-dose Iron Treatment in Non-anaemic Iron-deficient Women
Brief Title: Effectiveness of Low-dose Iron Treatment in Non-anaemic Iron-deficient Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Pierre-Alexandre Krayenbuehl, Clinical Professor, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LowdoseIron
Record Dates: First submitted 2020-11-09; First posted 2020-11-19 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Iron Deficiency (Without Anemia)
MeSH Terms: conditions — Iron Deficiencies | interventions — Iron, Dietary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iron-treatment group (Experimental)
  Interventions: Dietary Supplement: Eisen

INTERVENTIONS:
Dietary Supplement: Eisen — Treatment with low-dose iron in the form of tablets containing 6mg of iron. Treatment consists of twice-daily oral administration of iron-tablets for 8 weeks in total.

SUMMARY:
Iron deficiency is common in Switzerland and the main reason for anaemia. Nearly one in five premenopausal women suffers from iron deficiency. Low iron intake, reduced iron resorption or loss of blood are the main cause for iron deficiency. Symptoms of iron deficiency, for example fatigue, weakness, headache or exercise intolerance are primarily due to anaemia, but the same symptoms may also be present in non-anaemic patients with low serum ferritin. Consequently it is important to detect and treat non-anaemic iron deficiency. Common side effects of oral iron supplementation are primarily gastrointestinal symptoms like nausea, vomiting, diarrhea or abdominal pain. There is a positive correlation between appearance of gastrointestinal symptoms and administered iron dose. To date, only few studies have investigated effectiveness of low-dose iron supplementation in different target groups. The aim of this study is to investigate if low dose iron supplementation with 12mg iron per day for 8 weeks is sufficient to increase serum ferritin levels into a normal range in healthy premenopausal women suffering from non-anaemic iron deficiency

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Female gender
* Premenopausal
* Age > 18 years
* Regular menstrual cycle
* BMI in normal range (18-25 kg/m²)
* Serum-ferritin <30ng/ml
* No anaemia
* symptomatic iron deficiency in the past
* No intake of dietary supplements

Exclusion Criteria

* Intake of dietary supplements
* Pregnancy
* Hypermenorrhea
* Anaemia
* Serum-ferritin >30ng/ml
* BMI <18 kg/m² or >25 kg/m²
* chronic inflammatory diseases (e.g. colitis)
* Hypersensitivity to iron-supplements
* psychiatric disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Increase of serum ferritin concentration under iron supplementation | 8 weeks
  significant increase of serum-ferritin concentration after 8 weeks of low-dose iron-supplementation

SECONDARY OUTCOMES:
Side-effects of treatment | 8 weeks
  Adverse events will be assessed on a report form after 8 weeks
Serum hepcidin concentration | 8 weeks
  no increase in hepcidin-production during low-dose iron supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alexandre Krayenbühl, Principal Investigator — University of Zurich
Locations (1):
- Universitätsspital Zürich, Zurich, Switzerland

REFERENCES:
- [Derived] Simic S, Karczewski M, Klapdor S, Nowak A, Schubert M, Moretti D, Swinkels DW, Beuschlein F, Saleh L, Suter P, Krayenbuehl PA. Effectiveness of low-dose iron treatment in non-anaemic iron-deficient women: a prospective open-label single-arm trial. Swiss Med Wkly. 2023 May 25;153:40079. doi: 10.57187/smw.2023.40079. PMID 37229775